CLINICAL TRIAL: NCT06966700
Title: A Phase 3, Randomized, Open-label Study to Evaluate the Efficacy and Safety of Sac-TMT (Sacituzumab Tirumotecan, MK-2870) Followed by Carboplatin/Paclitaxel vs Chemotherapy, Both in Combination With Pembrolizumab as Neoadjuvant Therapy for High-Risk, Early-Stage, Triple-Negative Breast Cancer or Hormone Receptor-low Positive/Human Epidermal Growth Factor Receptor-2 Negative Breast Cancer
Brief Title: A Clinical Study of Sacituzumab Tirumotecan (Sac-TMT, MK-2870) in People With Breast Cancer (MK-2870-032)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2870-032; U1111-1316-7898 (Registry Identifier: UTN); 2024-520190-12-00 (Registry Identifier: EU CT); jRCT2031250231 (Registry Identifier: Japan Registry of Clinical Trial (jRCT))
Record Dates: First submitted 2025-05-04; First posted 2025-05-13 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Breast Neoplasms; Triple Negative Breast Neoplasms; HR Low-Positive/HER2-Negative Breast Neoplasms
Keywords: Programmed Cell Death-1 (PD1, PD-1); Programmed Cell Death 1 Ligand 1 (PDL1, PD-L1); Programmed Cell Death 1 Ligand 2 (PDL2, PD-L2)
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab; Carboplatin; Paclitaxel; Doxorubicin; Epirubicin; Cyclophosphamide; Capecitabine; olaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- sac-TMT (Experimental): Participants receive sacituzumab tirumotecan intravenously (IV) at a dose of 4 mg/kg every 2 weeks (Q2W) + IV pembrolizumab 200 mg every 3 weeks (Q3W), for 12 weeks; then receive IV pembrolizumab 200 mg Q3W and IV carboplatin area under the curve (AUC) 1.5 + IV paclitaxel 80 mg/m^2 once weekly, for 12 weeks. 3-6 weeks later, participants undergo surgery and optional radiation therapy, and receive IV pembrolizumab 400 mg once every 6 weeks or 200 mg Q3W for up to approximately 28 weeks. Additional adjuvant treatment of physician's choice (TPC) may be administered to participants with residual disease. TPC options are olaparib 300 mg oral twice daily (BID) for 1 year (participants with germline breast cancer susceptibility gene mutation (gBRCAm) only); capecitabine 1000-1250 mg/m^2 oral twice daily on days 1-14 and 22-35 each cycle for 4 six-week cycles; or doxorubicin 60mg/m^2 (or epirubicin 90 mg/m^2) IV infusion Q3W/Q2W + cyclophosphamide 600 mg/m^2 IV infusion Q3W/Q2W for 4 doses.
  Interventions: Biological: Sacituzumab tirumotecan; Biological: Pembrolizumab; Drug: Rescue Medication; Drug: Carboplatin; Drug: Paclitaxel; Drug: Doxorubicin; Drug: Epirubicin; Drug: Cyclophosphamide; Drug: Capecitabine; Drug: Olaparib
- Chemotherapy (Active Comparator): Participants receive IV carboplatin AUC 1.5 and paclitaxel 80 mg/m^2 once weekly, alongside pembrolizumab 200 mg Q3W, for 6 weeks; then receive IV pembrolizumab 200 mg Q3W alongside IV cyclophosphamide 600 mg/m^2 Q3W and either doxorubicin 60 mg/m^2 Q3W or epirubicin 90 mg/m^2 Q3W, for up to 12 weeks. 3-6 weeks later, participants undergo surgery and optional radiation therapy, and receive IV pembrolizumab 400 mg once every 6 weeks or 200 mg Q3W for up to approximately 28 weeks. Additional adjuvant TPC may be administered to participants with residual disease. TPC options are olaparib 300 mg oral BID for 1 year (participants with germline breast cancer susceptibility gene mutation (gBRCAm) only); or capecitabine 1000-1250 mg/m^2 oral BID on days 1-14 and 22-35 each cycle for 4 six-week cycles.
  Interventions: Biological: Pembrolizumab; Drug: Rescue Medication; Drug: Carboplatin; Drug: Paclitaxel; Drug: Doxorubicin; Drug: Epirubicin; Drug: Cyclophosphamide; Drug: Capecitabine; Drug: Olaparib

INTERVENTIONS:
Biological: Sacituzumab tirumotecan — IV infusion
  Other Names: Sac-TMT; MK-2870
  Arms: sac-TMT
Biological: Pembrolizumab — IV infusion
  Other Names: MK-3475; Keytruda®
Drug: Rescue Medication — Participants receive rescue medication at the investigators discretion, per approved product label. Recommended rescue medications are histamine -1 (H1) receptor agonist, histamine-2 (H2) receptor antagonist, acetaminophen or equivalent, dexamethasone or equivalent infusion, or steroid mouthwash (dexamethasone or equivalent).
Drug: Carboplatin — IV infusion
  Other Names: Paraplatin
Drug: Paclitaxel — IV infusion
  Other Names: Taxol; Onxol
Drug: Doxorubicin — IV infusion
  Other Names: ADRIAMYCIN®
Drug: Epirubicin — IV infusion
  Other Names: Ellence®
Drug: Cyclophosphamide — IV infusion
  Other Names: Cytophosphane
Drug: Capecitabine — Oral tablet
  Other Names: Xeloda®
Drug: Olaparib — Oral tablet
  Other Names: LYNPARZA®

SUMMARY:
Researchers are looking for new ways to treat types of breast cancer that are both:

* High-risk, which means the cancer may have a higher chance of getting worse or coming back after treatment
* Early-stage, which means the cancer is in the breast or the lymph nodes around the breast The 2 types of breast cancer in this study are triple-negative breast cancer (TNBC) and hormone receptor (HR)-low positive/human epidermal growth factor receptor-2 (HER2) negative breast cancer. These cancers have zero or a low amount of a protein called HER2 and other proteins that attach to the hormones estrogen or progesterone.

Sacituzumab tirumotecan (also known as sac-TMT or MK-2870), the study medicine, is a type of targeted therapy. A targeted therapy is a treatment that works to control how specific types of cancer cells grow and spread.

The main goals of this study are to learn if people who receive sac-TMT, pembrolizumab, and chemotherapy:

* Have fewer cancer cells found in the tumors and lymph nodes removed during surgery compared to those who receive only pembrolizumab and chemotherapy
* Live longer without the cancer growing, spreading, or coming back compared to people who receive only pembrolizumab with chemotherapy

ELIGIBILITY:
Inclusion Criteria:

The main inclusion criteria include but are not limited to the following:

* Has previously untreated high-risk, early-stage, non-metastatic (M0) breast cancer (BC), defined as any of the following combined primary tumor (T) and regional lymph node (N) staging per AJCC 8th edition criteria as assessed by the investigator based on radiological and/or clinical assessment:

  * cT1c, N1-N2
  * cT2, N0-N2
  * cT3, N0-N2
  * cT4a-d, N0-N2
* The participant must have a centrally confirmed diagnosis of BC that is triple-negative or HR-low+/HER2- (defined as estrogen receptor (ER)-low+ expression in 1% to 10% cells and HER2-), as by the most recent American Society of Clinical Oncology (ASCO)/College of American Pathologists (CAP) guidelines.
* Provides a core needle biopsy from the primary breast tumor at screening to the central laboratory.
* Has Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 performed within 28 days before treatment randomization.
* Demonstrates adequate organ function.

Exclusion Criteria:

The main exclusion criteria include but are not limited to the following:

* Metastatic (Stage IV) breast cancer or clinical node stage 3 (cN3) nodal involvement
* Has received any prior treatment, including radiation, systemic therapy,and/or definitive surgery for currently diagnosed breast cancer
* Has undergone excisional biopsy of the primary tumor, axillary lymph node dissection, and/or axillary sentinel lymph node biopsy prior to study treatment.
* Received prior systemic anticancer therapy including investigational agents within 4 weeks before randomization.
* Received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent, or with an agent directed to another stimulatory or coinhibitory T-cell receptor (eg, CTLA-4, OX- 40, CD137).
* Received prior treatment with a TROP2-targeted antibody-drug conjugate (ADC).
* Received prior treatment with a topoisomerase I inhibitor-containing ADC.
* Received a live or live-attenuated vaccine within 30 days before the first dose of study intervention.
* Known additional malignancy that is progressing or has required active treatment within the past 5 years.
* Uncontrolled systemic disease.
* History of (noninfectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2400 (Estimated)
Dates: Start 2025-06-30 (Actual); Primary Completion 2033-03-23 (Estimated); Study Completion 2034-12-29 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants with Pathological Complete Response (pCR) at the Time of Definitive Surgery | Up to approximately 30 weeks
  pCR (ypT0/Tis ypN0) is defined as the absence of residual invasive cancer on hematoxylin and eosin evaluation of the complete resected breast specimen and all sampled regional lymph nodes after completion of neoadjuvant systemic therapy per current American Joint Committee on Cancer (AJCC) staging criteria assessed by the local pathologist at the time of definitive surgery.
Event-Free Survival (EFS) | Up to approximately 92 months
  EFS is defined as the time from randomization to disease progression that precludes surgery, local or distant recurrence, or death due to any cause, whichever occurs first.

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to approximately 115 months
  OS is defined as the time from randomization to death due to any cause.
Percentage of Participants with pCR with No Ductal Carcinoma in Situ (pCR-no DCIS) at the Time of Definitive Surgery | Up to approximately 30 weeks
  pCR-no ductal carcinoma in situ (DCIS) (ypT0 ypN0) is defined as the absence of residual invasive and in situ cancer on hematoxylin and eosin evaluation of the complete resected breast specimen and all sampled regional lymph nodes after completion of neoadjuvant systemic therapy per current AJCC staging criteria assessed by the local pathologist at the time of definitive surgery.
Percentage of Participants with pCR at the Time of Definitive Surgery (High-risk, early-stage, TNBC subset) | Up to approximately 30 weeks
  pCR (ypT0/Tis ypN0) is defined as the absence of residual invasive cancer on hematoxylin and eosin evaluation of the complete resected breast specimen and all sampled regional lymph nodes after completion of neoadjuvant systemic therapy per current American Joint Committee on Cancer (AJCC) staging criteria assessed by the local pathologist at the time of definitive surgery. The pCR will be presented for the subset of participants who enrolled with high-risk, early-stage, TNBC.
Event-Free Survival (EFS) (High-risk, early-stage, TNBC subset) | Up to approximately 92 months
  EFS is defined as the time from randomization to disease progression that precludes surgery, local or distant recurrence, or death due to any cause, whichever occurs first. The EFS will be presented for the subset of participants who enrolled with high-risk, early-stage, TNBC.
Overall Survival (OS) (High-risk, early-stage, TNBC subset) | Up to approximately 115 months
  OS is defined as the time from randomization to death due to any cause.
Distant Progression or Distant Recurrence-Free Survival (DPDRFS) | Up to approximately 92 months
  DPDRFS is defined as the time from randomization to first distant progression or distant recurrence event as assessed by investigator, or death due to any cause, whichever occurs first.
Change from Baseline in European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30) Global Health Status-Quality of Life Score | Baseline and up to approximately 3 years
  The EORTC-QLQ-C30 is a 30-item questionnaire developed to assess the QoL of cancer patients. Participant responses to Item 30 (""How would you rate your overall quality of life during the past week?") is scored on a 7-point scale (1=Very Poor to 7=Excellent). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. A higher value indicates a better level of function. The change from baseline in EORTC QLQ-C30 Item 30 score will be reported.
Change from Baseline in EORTC QLQ-C30 Physical Functioning Score | Baseline and up to approximately 3 years
  The EORTC QLQ-C30 is a 30-item questionnaire to assess the overall quality of life of cancer patients. Participant responses to questions about their physical functioning are scored on a 4-point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. A higher score indicates a better level of physical functioning.
Change from Baseline in EORTC QLQ-C30 Role Functioning Score | Baseline and up to approximately 3 years
  The EORTC QLQ-C30 is a 30-item questionnaire to assess the overall quality of life of cancer patients. Participant responses to questions about their role functioning are scored on a 4-point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. A higher score indicates a better level of physical functioning.
Change from Baseline in EORTC QLQ-C30 Fatigue Score | Baseline and up to approximately 3 years
  The EORTC QLQ-C30 is a 30-item questionnaire to assess the overall quality of life of cancer patients. Participant responses to questions about their fatigue are scored on a 4-point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. A lower score indicates a better level of function.
Change from Baseline in EORTC QLQ Breast Cancer 42 (BR42) Systemic Therapy Side Effects Score | Baseline and up to approximately 3 years
  The EORTC QLQ-BR42 is a 42-item questionnaire to assess the overall quality of life of breast cancer patients. Participant responses to questions about their systemic therapy side effects are scored on a 4-point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. A lower score indicates a lower level of side effects.
Number of Participants Who Experience One or More Adverse Events (AEs) | Up to approximately 67 weeks
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Number of Participants Who Discontinue Study Treatment Due to an AE | Up to approximately 54 weeks
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (193):
- United States (38):
  - Banner MD Anderson Cancer Center ( Site 0066), Gilbert, Arizona
  - Roy and Patricia Disney Family Cancer Center ( Site 0055), Burbank, California
  - Providence Medical Foundation ( Site 0080), Fullerton, California
  - Hoag Memorial Hospital Presbyterian ( Site 0010), Newport Beach, California
  - Helios Clinical Research ( Site 0061), Whittier, California
  - Saint Joseph Hospital ( Site 0062), Denver, Colorado
  - Intermountain Health St. Mary's Regional Hospital ( Site 0054), Grand Junction, Colorado
  - Florida Cancer Specialists - South ( Site 7004), Fort Myers, Florida
  - Bioresearch Partner ( Site 0072), Hialeah, Florida
  - Florida Cancer Specialists - North ( Site 7002), St. Petersburg, Florida
  - Fort Wayne Medical Oncology and Hematology ( Site 0084), Fort Wayne, Indiana
  - Franciscan Health ( Site 0077), Indianapolis, Indiana
  - Ochsner Clinic Foundation ( Site 0021), New Orleans, Louisiana
  - Louisiana State University Health Sciences Shreveport ( Site 0053), Shreveport, Louisiana
  - New England Cancer Specialists ( Site 0051), Westbrook, Maine
  - Mercy Medical Center - Baltimore ( Site 0015), Baltimore, Maryland
  - Washington University Siteman Cancer Center ( Site 0031), St Louis, Missouri
  - Cancer Partners of Nebraska ( Site 0068), Lincoln, Nebraska
  - Renown Regional Medical Center ( Site 0041), Reno, Nevada
  - Rutgers Cancer Institute of New Jersey ( Site 0076), New Brunswick, New Jersey
  - Altru Health System ( Site 0057), Grand Forks, North Dakota
  - Good Samaritan Hospital-TriHealth Cancer institute ( Site 0027), Cincinnati, Ohio
  - Avera McKennan Hospital ( Site 0002), Sioux Falls, South Dakota
  - Avera Cancer Institute - Yankton ( Site 0089), Yankton, South Dakota
  - Tennessee Cancer Specialists ( Site 7001), Knoxville, Tennessee
  - Nashville General Hospital ( Site 0017), Nashville, Tennessee
  - Hendrick Medical Center ( Site 0009), Abilene, Texas
  - JPS Oncology and Infusion Center ( Site 0083), Fort Worth, Texas
  - Kelsey Research Foundation ( Site 0042), Houston, Texas
  - Kelsey-Seybold Clinic ( Site 0088), Houston, Texas
  - Oncology Consultants P.A. ( Site 0073), Houston, Texas
  - Texas Oncology - San Antonio ( Site 8004), San Antonio, Texas
  - Intermountain Medical Center ( Site 0074), Murray, Utah
  - Bon Secours Cancer Institute at St. Francis ( Site 0048), Midlothian, Virginia
  - Oncology and Hematology Associates of Southwest Virginia (BRCC) ( Site 8005), Roanoke, Virginia
  - Cancer Care Northwest ( Site 0003), Spokane, Washington
  - Northwest Medical Specialties, PLLC ( Site 0067), Tacoma, Washington
  - University of Wisconsin-Madison ( Site 0024), Madison, Wisconsin
- Argentina (8):
  - Instituto de Investigaciones Clinicas Mar del Plata ( Site 6008), Mar del Plata, Buenos Aires
  - Hospital Italiano de Buenos Aires-ginecology ( Site 6003), Buenos Aires, Buenos Aires F.D.
  - Centro de Educación Médica e Investigaciones clínicas "Dr. Norberto Quirno" (CEMIC) ( Site 6005), Buenos Aires, Buenos Aires F.D.
  - Fundacion Ars Medica ( Site 6004), San Salvador de Jujuy, Jujuy Province
  - Sanatorio Parque ( Site 6002), Rosario, Santa Fe Province
  - Clínica Mayo de Urgencias Médicas Cruz Blanca S.R.L ( Site 6006), San Miguel de Tucumán, Tucumán Province
  - Sanatorio Finochietto ( Site 6007), Buenos Aires
  - Sanatorio Allende - Nueva Córdoba ( Site 6000), Córdoba
- Australia (2):
  - Chris O'Brien Lifehouse ( Site 1206), Camperdown, New South Wales
  - Monash Health ( Site 1201), Clayton, Victoria
- Belgium (4):
  - Centre Hospitalier Universitaire de Liège - Domaine Universitaire du Sart Tilman ( Site 3204), Liège, Liege
  - AZORG Campus Aalst-Moorselbaan ( Site 3201), Aalst, Oost-Vlaanderen
  - UZ Gent ( Site 3202), Ghent, Oost-Vlaanderen
  - CHU UCL Namur/Site Sainte Elisabeth ( Site 3203), Namur
- Brazil (10):
  - PRONUTRIR ( Site 6120), Fortaleza, Ceará
  - Hospital Araújo Jorge ( Site 6100), Goiânia, Goiás
  - Liga Norte Riograndense Contra o Câncer ( Site 6111), Natal, Rio Grande do Norte
  - Associação Hospitalar Beneficente São Vicente de Paulo ( Site 6115), Passo Fundo, Rio Grande do Sul
  - Irmandade da Santa Casa de Misericórdia de Porto Alegre ( Site 6102), Porto Alegre, Rio Grande do Sul
  - Hospital São Lucas da PUCRS ( Site 6103), Porto Alegre, Rio Grande do Sul
  - Clínica de Oncologia Reichow ( Site 6112), Blumenau, Santa Catarina
  - Fundação Pio XII - Hospital de Câncer de Barretos ( Site 6108), Barretos, São Paulo
  - Hospital de Base de São José do Rio Preto ( Site 6101), São José do Rio Preto, São Paulo
  - INCA Hospital do Câncer III ( Site 6107), Rio de Janeiro
- Canada (5):
  - Health Sciences North ( Site 0234), Greater Sudbury, Ontario
  - Princess Margaret Cancer Centre ( Site 0208), Toronto, Ontario
  - Jewish General Hospital ( Site 0200), Montreal, Quebec
  - CHU de Quebec Universite Laval - Hopital du Saint-Sacrement ( Site 0203), Québec, Quebec
  - CIUSSS de l'Estrie-CHUS ( Site 0206), Sherbrooke, Quebec
- China (26):
  - Anhui Provincial Cancer Hospital ( Site 2234), Hefei, Anhui
  - Beijing Cancer Hospital ( Site 2201), Beijing, Beijing Municipality
  - The First Affiliated hospital of Xiamen University-Breast Surgery ( Site 2224), Xiamen, Fujian
  - Guangdong Maternity and Child Health Care Hospital ( Site 2251), Guangzhou, Guangdong
  - Jiangmen Center Hospital ( Site 2243), Jiangmen, Guangdong
  - Liuzhou People's Hospital ( Site 2259), Liuchow, Guangxi
  - Guangxi Medical University Affiliated Tumor Hospital ( Site 2223), Nanning, Guangxi
  - Harbin Medical University Cancer Hospital ( Site 2204), Haerbin, Heilongjiang
  - Henan Cancer Hospital ( Site 2238), Zhengzhou, Henan
  - Wuhan Union Hospital ( Site 2239), Wuhan, Hubei
  - Xiangya Hospital of Central South University ( Site 2225), Changsha, Hunan
  - Nanjing Drum Tower Hospital ( Site 2217), Nanjing, Jiangsu
  - Jiangsu Province Hospital ( Site 2216), Nanjing, Jiangsu
  - The Third Hospital Of Nanchang ( Site 2218), Nanchang, Jiangxi
  - The First Hospital Of Jilin University ( Site 2207), Changchun, Jilin
  - The First Affiliated Hospital of Xi'an Jiaotong University ( Site 2203), Xi'an, Shaanxi
  - Jinan Central Hospital ( Site 2249), Jinan, Shandong
  - Shandong Cancer Hospital ( Site 2205), Jinan, Shandong
  - Fudan University Shanghai Cancer Center ( Site 2209), Shanghai, Shanghai Municipality
  - Deyang City People's Hospital ( Site 2244), Deyang, Sichuan
  - The Second People's Hospital of Neijiang ( Site 2242), Neijiang, Sichuan
  - Xinjiang Medical University Cancer Hospital - Urumqi ( Site 2230), Ürümqi, Xinjiang
  - Yunnan Province Cancer Hospital ( Site 2226), Kunming, Yunnan
  - The Second Affiliated Hospital of Zhejiang University School of Medicine ( Site 2212), Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital ( Site 2211), Hangzhou, Zhejiang
  - Zhejiang Provincial People's Hospital ( Site 2215), Hangzhou, Zhejiang
- Colombia (6):
  - Instituto de Cancerología-Oncology ( Site 6302), Medellín, Antioquia
  - FUNDACION CTIC CENTRO DE TRATAMIENTO E INVESTIGACION SOBRE CANCER LUIS CARLOS SARMIENTO ANGULO ( Site 6311), Bogotá, Bogota D.C.
  - Clinica Colsanitas S.A, Sede Clínica Universitaria Colombia ( Site 6309), Bogotá, Bogota D.C.
  - IMAT S.A.S ( Site 6300), Montería, Departamento de Córdoba
  - Oncologos del Occidente ( Site 6303), Pereira, Risaralda Department
  - Fundación Valle del Lili ( Site 6308), Cali, Valle del Cauca Department
- Finland (3):
  - Oulun yliopistollinen sairaala ( Site 3603), Oulu, North Ostrobothnia
  - Tampereen ylipistollinen sairaala ( Site 3601), Tampere, Pirkanmaa
  - Helsinki University Hospital - Comprehensive Cancer Center (HYKS - Syöpäkeskus) ( Site 3600), Helsinki, Uusimaa
- France (5):
  - Centre Georges Francois Leclerc ( Site 3902), Dijon, Bourgogne-Franche-Comté
  - Centre de Cancerologie du Grand Montpellier ( Site 3910), Montpellier, Herault
  - Centre Eugène Marquis Rennes - Centre de Lutte Contre le Cancer-Medical Oncology ( Site 3900), Rennes, Ille-et-Vilaine
  - CHU d'Amiens-Picardie - Hôpital Sud ( Site 3908), Amiens, Somme
  - HENRI MONDOR HOSPITAL ( Site 3904), Créteil, Val-de-Marne
- Guatemala (5):
  - MEDI-K ( Site 6400), Guatemala City
  - CELAN,S.A ( Site 6401), Guatemala City
  - INTEGRA Cancer Institute ( Site 6404), Guatemala City
  - Onco Go, S.A ( Site 6402), Guatemala City
  - Asociacion Española de Beneficencia ( Site 6403), Guatemala City
- Hong Kong (3):
  - Hong Kong United Oncology Centre ( Site 1304), Jordan
  - Queen Mary Hospital ( Site 1300), Pokfulam
  - Prince of Wales Hospital ( Site 1301), Shatin
- Bacs-Kiskun Varmegyei Oktatokorhaz-Onkoradiologiai Kozpont ( Site 4207), Kecskemét, Bács-Kiskun county, Hungary
- Israel (4):
  - Rambam Health Care Campus ( Site 4400), Haifa
  - Meir Medical Center. ( Site 4403), Kfar Saba
  - Sheba Medical Center ( Site 4401), Ramat Gan
  - Yitzhak Shamir Medical Center. ( Site 4404), Ẕerifin
- Japan (19):
  - Nagoya City University Hospital ( Site 2310), Nagoya, Aichi-ken
  - National Hospital Organization Hokkaido Cancer Center ( Site 2300), Sapporo, Hokkaido
  - Kanagawa Cancer Center ( Site 2308), Yokohama, Kanagawa
  - Mie University Hospital ( Site 2312), Tsu, Mie-ken
  - Kansai Medical University Hospital ( Site 2317), Hirakata, Osaka
  - Kindai University Hospital ( Site 2316), Sakai, Osaka
  - The University of Osaka Hospital ( Site 2314), Suita, Osaka
  - Shizuoka Cancer Center ( Site 2309), Sunto-gun, Shizuoka
  - National Cancer Center Hospital ( Site 2305), Chūō, Tokyo
  - Toranomon Hospital ( Site 2307), Minato, Tokyo
  - Showa Medical University Hospital ( Site 2306), Shinagawa, Tokyo
  - Akita University Hospital ( Site 2302), Akita
  - Chiba Cancer Center ( Site 2303), Chiba
  - Fukushima Medical University Hospital ( Site 2301), Fukushima
  - Hiroshima City Hiroshima Citizens Hospital ( Site 2318), Hiroshima
  - Kumamoto Shinto General Hospital ( Site 2322), Kumamoto
  - Kyoto University Hospital ( Site 2313), Kyoto
  - Nakagami Hospital ( Site 2323), Okinawa
  - National Hospital Organization Osaka National Hospital ( Site 2315), Osaka
- Malaysia (4):
  - Hospital Pulau Pinang ( Site 1502), George Town, Pulau Pinang
  - National Cancer Institute ( Site 1501), Putrajaya, Putrajaya
  - Sarawak General Hospital ( Site 1504), Kuching, Sarawak
  - Pantai Hospital Kuala Lumpur ( Site 1500), Kuala Lumpur
- Peru (3):
  - Instituto Regional de Enfermedades Neoplasicas del Centro (IREN CENTRO) ( Site 6605), Concepción, Departamento de Junín
  - IPOR Instituto Peruano de Oncología & Radioterapia ( Site 6600), Lima
  - Oncosalud ( Site 6603), Lima
- Poland (3):
  - Centrum Onkologii im. Prof. Franciszka Lukaszczyka ( Site 4616), Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie - Panstwowy Instytut Badawczy w Warszawie ( Site 4609), Warsaw, Masovian Voivodeship
  - Szpital Kliniczny Ministerstwa Spraw Wewnętrznych i Administracji z Warmińsko-Mazurskim Centrum Onko ( Site 4614), Olsztyn, Warmian-Masurian Voivodeship
- Portugal (2):
  - Unidade Local de Saude Lisboa Ocidental - Hospital de São Francisco Xavier ( Site 4702), Lisbon, Lisbon District
  - Hospital de Cascais Doutor José de Almeida ( Site 4700), Lisbon
- National Cancer Centre Singapore ( Site 1700), Singapore, Central Singapore, Singapore
- South Africa (5):
  - CANCERCARE LANGENHOVEN DRIVE ONCOLOGY CENTRE ( Site 4907), Port Elizabeth, Eastern Cape
  - Wits Clinical Research ( Site 4903), Johannesburg, Gauteng
  - LIFE GROENKLOOF-Mary Potter Cancer Centre ( Site 4901), Pretoria, Gauteng
  - Sandton Oncology Medical Group (Pty) Ltd ( Site 4900), Sandton, Gauteng
  - Cancercare Rondebosch Oncology ( Site 4906), Cape Town, Western Cape
- South Korea (8):
  - National Cancer Center ( Site 1800), Goyang-si, Kyonggi-do
  - Seoul National University Bundang Hospital ( Site 1801), Kyonggi-do, Kyonggi-do
  - Kyungpook National University Chilgok Hospital ( Site 1805), Taegu, Taegu-Kwangyokshi
  - Seoul National University Hospital ( Site 1806), Seoul
  - Severance Hospital Yonsei University Health System ( Site 1804), Seoul
  - Asan Medical Center ( Site 1803), Seoul
  - Samsung Medical Center ( Site 1807), Seoul
  - The Catholic University of Korea. Seoul St. Mary s Hospital ( Site 1802), Seoul
- Spain (10):
  - Institut Català d'Oncologia - L'Hospitalet ( Site 5001), L'Hospitalet de Llobregat, Barcelona
  - Hospital de Basurto ( Site 5007), Bilbao, Bizkaia
  - Complejo asistencial universitario de Salamanca ( Site 5000), Salamanca, Castille and León
  - HOSPITAL UNIVERSITARIO DE JAEN ( Site 5003), Jaén, Jaen
  - CHUS - Hospital Clinico Universitario ( Site 5006), Santiago de Compostela, La Coruna
  - HOSPITAL UNIVERSITARIO QUIRONSALUD MADRID ( Site 5004), Pozuelo de Alarcón, Madrid
  - Hospital General de Valencia ( Site 5008), Valencia, Valenciana, Comunitat
  - Parc de Salut Mar - Hospital del Mar ( Site 5005), Barcelona
  - Hospital Beata María Ana ( Site 5010), Madrid
  - Hospital Universitario Virgen Macarena ( Site 5002), Seville
- Sweden (4):
  - Skånes Universitetssjukhus Malmö ( Site 3802), Malmo, Skåne County
  - Karolinska Universitetssjukhuset Solna ( Site 3800), Stockholm, Stockholm County
  - Akademiska sjukhuset ( Site 3801), Uppsala, Uppsala County
  - Södra Älvsborgs Sjukhus Borås ( Site 3804), Borås, Västra Götaland County
- Taiwan (5):
  - Taichung Veterans General Hospital ( Site 1904), Taichung
  - National Taiwan University Hospital ( Site 1900), Taipei
  - MacKay Memorial Hospital ( Site 1903), Taipei
  - National Taiwan University Cancer Center (NTUCC) ( Site 1901), Taipei
  - Chang Gung Medical Foundation-Linkou Branch ( Site 1906), Taoyuan District
- Faculty of Medicine Siriraj Hospital ( Site 2000), Bangkok, Bangkok, Thailand
- Ukraine (5):
  - COMMUNAL NONPROFIT ENTERPRISE "CLINICAL CENTER OF ONCOLOGY, HEMATOLOGY, TRANSPLANTOLOGY AND PALLIATI ( Site 5207), Cherkasy, Cherkasy Oblast
  - Municipal Enterprise "Bukovinian сlinical oncology сenter" ( Site 5208), Chernivtsi, Chernivetska Oblast
  - CNCE Precarpathian Clinical Oncologic Center ( Site 5201), Ivano-Frankivsk, Ivano-Frankivsk Oblast
  - CNE Regional clinical oncology center of Kirovograd regional Council ( Site 5203), Kropyvnytsky, Kirovohrad Oblast
  - Shalimov Institute of Surgery and Transplantation ( Site 5210), Kyiv
- United Kingdom (3):
  - Ninewells Hospital and Medical School ( Site 5300), Dundee, Dundee City
  - Huddersfield Royal Infirmary ( Site 5313), Huddersfield, England
  - St Bartholomew s Hospital ( Site 5302), London, London, City of

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/